CLINICAL TRIAL: NCT03191084
Title: Examine the Feasibility of a Standardized Field Test for Marijuana Impairment: Laboratory Evaluations
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Highway Traffic Safety Administration (NHTSA) (U.S. Federal Agency); Hartford Hospital (Other); Montana State University (Other); Maastricht University (Other); The Mind Research Network (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Godfrey Pearlson, Principal Investigator, Yale University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: 2000021338; DTNH2216C00022 (Other: Department of Transportation, (U.S.))
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Marijuana Impairment
Keywords: marijuana; THC; cannabis; driving; impairment; intoxication
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol; nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regular Users (Experimental): People who use marijuana regularly will be given a low dose THC marijuana, high dose THC marijuana and placebo marijuana, in a randomized order, at the five study visits.
  Interventions: Drug: Low Dose THC Marijuana; Drug: High Dose THC Marijuana; Drug: Placebo Marijuana
- Occasional Users (Experimental): People who use marijuana occasionally will be given a low dose THC marijuana, high dose THC marijuana and placebo marijuana, in a randomized order, at the five study visits.
  Interventions: Drug: Low Dose THC Marijuana; Drug: High Dose THC Marijuana; Drug: Placebo Marijuana

INTERVENTIONS:
Drug: Low Dose THC Marijuana — Dosing via vaporized marijuana using a lower concentration of THC, participants receive this dose on two of the five study visits.
  Other Names: THC, Cannabis
Drug: High Dose THC Marijuana — Dosing via vaporized marijuana using a higher concentration of THC, participants receive this dose on two of the five study visits.
  Other Names: THC, Cannabis
Drug: Placebo Marijuana — Dosing via vaporized marijuana with no THC, participants receive this dose on one of the five study visits.
  Other Names: THC, Cannabis

SUMMARY:
Marijuana is one of the most widely used substances. This study will characterize the persistence of cannabis' (CNB's) acute effects on cognitive test performance and simulated driving over a several hour time period. The data obtained from simulated driving, cognitive tests, and biological assays of THC will be used in analyses aimed at identifying what tests or combination of tests predict both recent use and driving impairment risk.

Eligible participants will undergo a full day screening visit, if still eligible they will come to Hartford Hospital in Hartford, Connecticut to take part in the full study. Participation requires overnight stays between each of the five study visits. On each of the study days participants are dosed with either a low dose of THC marijuana, a high dose of THC marijuana or placebo marijuana, (the low and high doses are repeated once each, order in which the study drug is given is double blind and chosen at random.)

DETAILED DESCRIPTION:
This responds to NHTSA's request with a proposal to increase our understanding of smoked cannabis' (CNB's) acute effects on cognition and simulated driving performance, the persistence of these deficits over the hours after use, and the influence of prior experience with CNB on these effects. The project also will link an extensive literature on CNB's effects on laboratory cognitive tests to simulated driving performance for the first time, providing a crucial validation of CNB's neurofunctional effects identifying maximally relevant candidate measures for field sobriety tests. To this goal, the proposed study was based upon a careful and thorough review of the scientific literature describing CNB effects on cognitive test performance and driving, as well as current state-of-knowledge on the sensitivity of biological assays for identifying recent CNB use. The study will carefully characterize the persistence of CNB's acute effects on cognitive test performance and driving over a several-hour time span. This will allow us to identify the point at which any effects of CNB intoxication on cognitive tests and driving performance cannot be distinguished from normal, i.e., the first step towards establishing standards for legal and social policy. The data obtained from simulated driving, cognitive tests, and biological assays of THC will be used in analyses aimed at identifying what tests or combination of tests predict both recent use and driving impairment risk.

Participants

ELIGIBILITY:
Inclusion Criteria:

* Must have a current driver's license
* Have used marijuana before
* Right handed

Exclusion Criteria:

* Females who are pregnant or breast feeding
* Any serious medical, or neurological disorder
* Any psychiatric disorder
* No major head traumas

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Marijuana induced performance changes on Cogstate 1-back/2-back task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours; 4.5 hours; 6.5 hours
  The Cogstate 1-back/2-back task assesses working memory, it will be administered prior to dosing and at various time points after dosing.
Marijuana induced performance changes on Cogstate Card Learning. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours; 4.5 hours; 6.5 hours
  The Cogstate Card Learning task assesses visual memory, it will be administered prior to dosing and at various time points after dosing.
Marijuana induced performance changes on Cogstate Groton Maze Learning task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours; 4.5 hours; 6.5 hours
  The Cogstate Groton Maze Learning task assesses spatial learning and memory, it will be administered prior to dosing and at various time points after dosing.
Marijuana induced performance changes on Cogstate Social/Emotional Cognition task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours; 4.5 hours; 6.5 hours
  The Cogstate Social/Emotional Cognition task assesses emotional processing, it will be administered prior to dosing and at various time points after dosing.
Marijuana induced performance changes on Alertmeter. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours; 4.5 hours; 6.5 hours
  The Alertmeter task assess visual judgment and alertness, it will be administered prior to dosing and at various time points after dosing.
Marijuana induced performance changes on the Time Estimation Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours; 4.5 hours; 6.5 hours
  The Time Estimation Task assesses timing, it will be administered prior to dosing and at various time points after dosing.
Marijuana induced performance changes on the Stop Signal Reaction Time task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours; 4.5 hours; 6.5 hours
  The Stop Signal Reaction Time Task assesses inhibitory processing, it will be administered prior to dosing and at various time points after dosing.
Marijuana induced performance changes on the Critical Tracking Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours; 4.5 hours; 6.5 hours
  The Critical Tracking Task assesses hand eye coordination and visuomotor tracking, it will be administered prior to dosing and at various time points after dosing.
Marijuana induced performance changes on the ANAM Pursuit Tracking Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours; 4.5 hours; 6.5 hours
  The ANAM Pursuit Tracking Task assesses hand eye coordination, it will be administered prior to dosing and at various time points after dosing.
Marijuana induced performance changes on the Finger to Nose Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours; 4.5 hours; 6.5 hours
  The Finger to Nose Task assesses general motor coordination, it will be administered prior to dosing and at various time points after dosing.
Marijuana induced performance changes on the One Leg Stand Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours; 4.5 hours; 6.5 hours
  The One Leg Stand Task assesses general motor coordination, it will be administered prior to dosing and at various time points after dosing.
Marijuana induced performance changes on the Line Walking/Months Backwards Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours; 4.5 hours; 6.5 hours
  The Line Walking/Months Backwards Task assesses general motor coordination plus distraction, it will be administered prior to dosing and at various time points after dosing.
Marijuana induced performance changes on the Time Reproduction Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours; 4.5 hours; 6.5 hours
  The Time Reproduction Task assesses general motor coordination plus timing, it will be administered prior to dosing and at various time points after dosing.

SECONDARY OUTCOMES:
Change in concentration of THC/metabolites in blood samples. | Baseline and post drug administration at: 5 min, 20 min, 1 hr 10 min, 1 hr 45 min, 2 hrs 30 min, 4 hrs, and 6 hrs 30 min.
  Blood samples with be collected at 8 times throughout each day to assess for changes of THC and its metabolite levels.
Change in concentration of THC/metabolites in oral fluid tested using Draeger Drug Detection Kits. | Baseline and post drug administration at: 5 min, 20 min, 1 hr 10 min, 1 hr 45 min, 2 hrs 30 min, 4 hrs, and 6 hrs 30 min.
  Oral fluid samples with be collected at 8 times throughout each day to assess for changes of THC and its metabolite levels.
Change in concentration of THC/metabolites in oral fluid tested using Quantisal Oral Fluid Collection devices. | Baseline and post drug administration at: 5 min, 20 min, 1 hr 10 min, 1 hr 45 min, 2 hrs 30 min, 4 hrs, and 6 hrs 30 min.
  Oral fluid samples with be collected at 8 times throughout each day to assess for changes of THC and its metabolite levels.
Change in performance on simulated driving Road Tracking Task. | Post drug administration at: 1 hour, 3 hours and 5 hours
  The Road Tracking Task measures operational control of the vehicle. Operational control is measured by standard deviation of lane position from the center point of the lane.
Change in performance on simulated driving Car Following Task. | Post drug administration at: 1 hour, 3 hours and 5 hours
  The Car Following Task measures tactical control of the vehicle. Tactical control of the vehicle is measured by following distance from a lead vehicle.
Change in performance on simulated driving Gap Acceptance Task. | Post drug administration at: 1 hour, 3 hours and 5 hours
  The Gap Acceptance Task measures strategic control of the vehicle. Strategic control of the vehicle is measured by size of headway gaps that the participant chooses in pulling out into oncoming traffic to overtake a stopped car.

CONTACTS AND LOCATIONS:
Locations (1):
- Olin Neuropsychiatry Research Center, Hartford, Connecticut, United States